CLINICAL TRIAL: NCT03616587
Title: A Phase 1 Dose Escalation and Expansion Study of AZD9833 Alone or in Combination in Women With ER-positive, HER2-negative Advanced Breast Cancer (SERENA-1)
Brief Title: Study of AZD9833 Alone or in Combination in Women With Advanced Breast Cancer.
Acronym: SERENA-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8530C00001; 138396 (Registry Identifier: IND); 2023-506890-37-00 (Registry Identifier: CTIS); 2018-000667-92 (EudraCT Number)
Record Dates: First submitted 2018-07-06; First posted 2018-08-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: ER+ HER2- Advanced Breast Cancer
Keywords: Breast Cancer; Phase 1; Safety; Tolerability; Pharmacokinetics; ER Positive; HER2 Negative; Advanced Breast Cancer; Camizestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — AZD9833; palbociclib; Everolimus; abemaciclib; capivasertib; ribociclib; Anastrozole

STUDY DESIGN:
Intervention Model Description: Dose escalation and expansion, first-in-human study to evaluate safety and tolerability of AZD9833 alone (Parts A and B) or in combination with palbociclib (Parts C and D) or with everolimus (Parts E and F) or with abemaciclib (±anastrozole) (Parts G and H) or with capivasertib (Parts I and J) or with ribociclib (±anastrozole) (Parts K and L) or with anastrozole (Parts M and N) in women with endocrine-resistant ER+ HER2- breast cancer not amenable to curative treatment.
  Parts A, C, E, G, I, K, and M allow for dose escalation and/or de-escalation of AZD9833 alone or in combination with palbociclib, everolimus, abemaciclib (± anastrozole), capivasertib, ribociclib (± anastrozole) or anastrozole.
  Based on the findings in dose escalation, the expansions (Parts B, D, F, H, J, L, N) will further investigate selected doses of AZD9833, alone or in combination with palbociclib, everolimus ,abemaciclib (±anastrozole), capivasertib ,ribociclib(±anastrozole) and anastrozole.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- AZD9833 monotherapy dose escalation (Experimental)
  Interventions: Drug: AZD9833
- AZD9833 monotherapy dose expansion (Experimental)
  Interventions: Drug: AZD9833
- AZD9833 with palbociclib dose escalation (Experimental)
  Interventions: Drug: AZD9833 with palbociclib
- AZD9833 with palbociclib dose expansion (Experimental)
  Interventions: Drug: AZD9833 with palbociclib
- AZD9833 with everolimus dose expansion (Experimental)
  Interventions: Drug: AZD9833 with everolimus
- AZD9833 with everolimus dose escalation (Experimental)
  Interventions: Drug: AZD9833 with everolimus
- AZD9833 with abemaciclib (± anastrozole) dose escalation (Experimental)
  Interventions: Drug: AZD9833 with abemaciclib
- AZD9833 with abemaciclib (± anastrozole)dose expansion (Experimental)
  Interventions: Drug: AZD9833 with abemaciclib
- AZD9833 with capivasertib dose escalation (Experimental)
  Interventions: Drug: AZD9833 with capivasertib
- AZD9833 with capivasertib dose expansion (Experimental)
  Interventions: Drug: AZD9833 with capivasertib
- AZD9833 with ribociclib (± anastrozole) dose escalation (Experimental)
  Interventions: Drug: AZD9833 with ribociclib
- AZD9833 with ribociclib (± anastrozole) dose expansion (Experimental)
  Interventions: Drug: AZD9833 with ribociclib
- AZD9833 with anastrozole dose escalation (Experimental)
  Interventions: Drug: AZD9833 with anastrozole
- AZD9833 with anastrozole dose expansion (Experimental)
  Interventions: Drug: AZD9833 with anastrozole

INTERVENTIONS:
Drug: AZD9833 — Part A: AZD9833 monotherapy dose escalation.
  Arms: AZD9833 monotherapy dose escalation
Drug: AZD9833 — Part B: AZD9833 monotherapy expansion.
  Arms: AZD9833 monotherapy dose expansion
Drug: AZD9833 with palbociclib — Part C: AZD9833 in combination with palbociclib dose escalation
  Arms: AZD9833 with palbociclib dose escalation
Drug: AZD9833 with palbociclib — Part D: AZD9833 in combination with palbociclib expansion
  Arms: AZD9833 with palbociclib dose expansion
Drug: AZD9833 with everolimus — Part E: AZD9833 in combination with everolimus dose escalation
  Arms: AZD9833 with everolimus dose escalation
Drug: AZD9833 with everolimus — Part F: AZD9833 in combination with everolimus dose expansion
  Arms: AZD9833 with everolimus dose expansion
Drug: AZD9833 with abemaciclib — Part G: AZD9833 in combination with abemaciclib (± anastrozole) dose escalation
  Arms: AZD9833 with abemaciclib (± anastrozole) dose escalation
Drug: AZD9833 with abemaciclib — Part H: AZD9833 in combination with abemaciclib (± anastrozole) dose expansion
  Arms: AZD9833 with abemaciclib (± anastrozole)dose expansion
Drug: AZD9833 with capivasertib — Part I: AZD9833 in combination with capivasertib dose escalation
  Arms: AZD9833 with capivasertib dose escalation
Drug: AZD9833 with capivasertib — Part J: AZD9833 in combination with capivasertib dose expansion
  Arms: AZD9833 with capivasertib dose expansion
Drug: AZD9833 with ribociclib — Part K: AZD9833 in combination with ribociclib (± anastrozole) dose escalation
  Arms: AZD9833 with ribociclib (± anastrozole) dose escalation
Drug: AZD9833 with ribociclib — Part L: AZD9833 in combination with ribociclib (± anastrozole) dose expansion
  Arms: AZD9833 with ribociclib (± anastrozole) dose expansion
Drug: AZD9833 with anastrozole — Part M: AZD9833 in combination with anastrozole dose escalation
  Arms: AZD9833 with anastrozole dose escalation
Drug: AZD9833 with anastrozole — Part N: AZD9833 in combination with anastrozole dose expansion
  Arms: AZD9833 with anastrozole dose expansion

SUMMARY:
A Phase 1 Dose Escalation and Expansion Study of AZD9833 Alone or in Combination in Women with ER Positive, HER2 Negative Advanced Breast Cancer (SERENA-1)

DETAILED DESCRIPTION:
This is a multicentre dose escalation and expansion, first-in-human study designed to evaluate the safety and tolerability of AZD9833, alone (Parts A and B), or in combination with palbociclib (Parts C and D), or in combination with everolimus (Parts E and F), or in combination with abemaciclib (± anastrozole) (Parts G and H), or in combination with capivasertib (Parts I and J), or in combination with ribociclib (± anastrozole) (Parts K and L), or in combination with anastrozole (Parts M and N) in women with endocrine-resistant ER+ HER2- breast cancer that is not amenable to treatment with curative intent.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. >= 18 years
3. Any menopausal status:

   1. Pre-menopausal women must have commenced treatment with an LHRH agonist at least 4 weeks prior to starting AZD9833 (± combination IMP(s)) and must be willing to continue to receive LHRH agonist therapy for the duration of the study
   2. Post-menopausal defined according to standard criteria in the protocol.
4. Histological or cytological confirmation of adenocarcinoma of the breast
5. Documented positive oestrogen receptor status of primary or metastatic tumour tissue, according to the local laboratory parameters.HER-2 negative.
6. Metastatic disease or locoregionally recurrent disease which is refractory or intolerant to existing therapy(ies) known to provide clinical benefit
7. Metastatic or locoregionally recurrent disease and radiological or objective evidence of progression on or after the last systemic therapy prior to starting IMP
8. Prior chemotherapy, endocrine therapy and other therapy as follows:

   1. No more than 2 lines of chemotherapy for advanced disease
   2. Recurrence or progression on at least one line of endocrine therapy in the advanced/metastatic disease setting
   3. There is no limit on the number of lines of prior endocrine therapies
   4. Prior treatment with CDK4/6 inhibitors is permitted
9. Women of childbearing potential must agree to use a highly effective contraceptive measure, must not be breast feeding, and must have a negative pregnancy test prior to the start of dosing.
10. At least one lesion (measurable and/or non-measurable, as per RECIST 1.1 that can be accurately assessed at baseline and is suitable for repeated assessment by CT, MRI, or plain X-ray; or clinical examination. Blastic-only lesions in bone are not considered assessable.
11. ECOG/ WHO performance status 0 to 1, with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks Inclusion criteria for the paired tumour biopsy research:

    Inclusion criteria for the paired tumour biopsy research
12. Disease suitable for paired baseline and on-study tumour biopsies
13. Washout from prior fulvestrant: 6 months
14. Washout from prior tamoxifen: 4 months
15. Signed written informed consent for tumour biopsies

Exclusion Criteria

1. Intervention with any of the following

   1. Any cytotoxic chemotherapy, investigational agents/other anti-cancer drugs for the treatment of advanced breast cancer from a previous treatment regimen or clinical study within 14 days of the first dose of IMP
   2. Concomitant medications or herbal supplements known to be strong inhibitors/inducers of cytochrome P450 (CYP) 3A4/5, sensitive CYP2B6 substrates, and drugs which are sensitive substrates of CYP2C9 and/or CYP2C19, and which have a narrow therapeutic index. In addition: Parts E and F will exclude the concomitant use of moderate CYP3A4 and/or Pgp inhibitors; Parts G H, I, J, K and L will exclude the concomitant use of moderate CYP3A4/5 inhibitors and inducers; Parts I and J will exclude concomitant use of sensitive substrates of CYP3A4 and/or CYP2D6 with a narrow therapeutic index."
   3. Drugs known to prolong QT and known risk of Torsades de Pointes
   4. Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of IMP, except patients receiving radiotherapy to more than 30% of the bone marrow/a wide field of radiation within 4 weeks of the first dose of IMP
   5. Major surgical procedure/significant traumatic injury, as judged by the investigator, within 4 weeks of the first dose of IMP, or an anticipated need for major surgery and/or any surgery requiring general anaesthesia during the study.
2. Any unresolved toxicities from prior therapy > CTCAE Grade 1 at the time of starting IMP, with the exception of alopecia.
3. Presence of life-threatening metastatic visceral disease, as judged by the investigator, uncontrolled CNS metastatic disease. Patients with spinal cord compression and/or brain metastases may be enrolled if definitively treated (eg, surgery or radiotherapy) and stable off steroids for at least 4 weeks prior to start of IMP
4. Past medical history of ILD (Parts E, F, K and L only)
5. Currently symptomatic radiotherapy-induced pneumonitis (Parts E, F, K and L only)
6. Evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C, and human immunodeficiency virus (HIV)
7. Any of the following cardiac criteria

   1. Mean resting QTcF >470 msec obtained from a triplicate ECG (≥450 msec for Parts K and L)
   2. Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG (eg, complete left bundle branch block, second- and third-degree heart block), or clinically significant sinus pause. Patients with controlled atrial fibrillation can be enrolled c) Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as symptomatic heart failure, hypokalaemia, congenital long QT syndrome, immediate family history of long QT syndrome, or unexplained sudden death at <40 years of age. Hypertrophic cardiomyopathy and clinically significant stenotic valve disease

   (d) LVEF <50% and/or experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, unstable angina pectoris, congestive heart failure NYHA Grade ≥2, cerebrovascular accident, or transient ischaemic attack.

   (e) Uncontrolled hypertension. Hypertensive patients may be eligible but blood pressure must be adequately controlled at baseline.

   (f) Uncontrolled hypotension - SBP <90 mmHg and/or DBP <50 mmHg for parts I &J
8. Inadequate bone marrow reserve/organ function as demonstrated by any of the following lab values

   1. ANC <1.5 × 109/L
   2. Platelet count <100 × 109/L
   3. Haemoglobin <90 g/L
   4. ALT >2.5 × ULN
   5. AST >2.5 × ULN
   6. TBL >1.5 × ULN or >3 × ULN in the presence of documented Gilbert's Syndrome
   7. GFR <50 mL/min
9. Clinically significant abnormalities of glucose metabolism, as defined by any of the following at screening (Parts I and J only):

   1. Patients with diabetes mellitus type I or diabetes mellitus type II requiring insulin treatment.
   2. HbA1c ≥8.0% (63.9 mmol/mol).

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pre-menopausal or Post-menopausal women
Enrollment: 396 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2027-06-24 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with dose-limiting toxicity, as defined in the protocol. | Minimum observation period 28 days on treatment.
  Dose-limiting toxicity as described in the protocol that is not related to disease progression, intercurrent illness or concomitant medications and that, despite optimal therapeutic intervention, meets protocol-defined criteria.
The number of subjects with treatment-related adverse events as assessed by CTCAE v4.03. | Minimum observation period 28 days on treatment, and will continue until the subject is off the study (approximately 1 year).
  Data will include clinical observations, ECG parameters, clinical chemistry and haematology and vital signs assessed as the number of subjects with treatment-related adverse events assessed by CTCAE v4.03.

SECONDARY OUTCOMES:
Objective Response Rate | Weeks 8, 16 and 24 and then every 12 weeks (weeks 36, 48 and 60) until the end of the study (approximately 1 year).
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Duration of Response | Weeks 8, 16 and 24 and then every 12 weeks (weeks 36, 48 and 60) until the end of the study (approximately 1 year).
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Clinical benefit rate at 24 weeks | Up to 24 weeks
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Percentage Change in Tumour Size | Weeks 8, 16 and 24 and then every 12 weeks (weeks 36, 48 and 60) until the end of the study (approximately 1 year).
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Progression Free Survival | Weeks 8, 16 and 24 and then every 12 weeks (weeks 36, 48 and 60) until the end of the study (approximately 1 year).
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Maximum Observed Plasma Concentration (Cmax) of AZD9833 alone or in combination with Palbociclib, Everolimus, Abemaciclib, Capivasertib, Ribociclib or Anastrozole | At predefined intervals throughout the AZD9833 treatment period (approximately 16 weeks )
  Blood samples will be collected to assess plasma concentrations of AZD9833 alone or in combination with Palbociclib, Everolimus, Abemaciclib, Capivasertib, Ribociclib or Anastrozole at a series of timepoints to derive Cmax
Time to observed Cmax (Tmax) for AZD9833 alone or in combination with Palbociclib, Everolimus, Abemaciclib, Capivasertib, Ribociclib or Anastrozole | At predefined intervals throughout the AZD9833 treatment period (approximately 16 weeks )
  Blood samples will be collected to assess plasma concentrations of AZD9833 alone or in combination with Palbociclib, Everolimus, Abemaciclib, Capivasertib, Ribociclib or Anastrozole at a series of timepoints to derive Tmax
Area under the plasma concentration-time curve (AUC) for AZD9833 alone or in combination with Palbociclib, Everolimus, Abemaciclib, Capivasertib, Ribociclib or Anastrozole | At predefined intervals throughout the AZD9833 treatment period (approximately 16 weeks )
  Blood samples will be collected to assess plasma concentrations of AZD9833 alone or in combination with Palbociclib, Everolimus, Abemaciclib, Capivasertib, Ribociclib or Anastrozole at a series of timepoints to derive AUC
Renal clearance (CLR) for AZD9833 | At predefined intervals throughout the AZD9833 treatment period (approximately 16 weeks )
  Urine samples will be collected to assess urine concentrations of AZD9833 at a series of timepoints to derive renal clearance
Assessment of biomarker changes | At pre-defined time intervals throughout the AZD9833 treatment period and at discontinuation. (approximately 1 year)
  Tumour samples will be collected to assess biomarker changes of estrogen receptor (ER), progesterone receptor (PgR) and Ki67 protein at a series of timepoints to derive AZD9833 activity in tumour cells.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Baird, MD PhD FRCP, Principal Investigator — Breast Cancer Research Unit, University of Cambridge; Justin Lindemann, MBChB MBA, Study Director — AstraZeneca
Locations (14):
- United States (5):
  - Research Site, Aurora, Colorado
  - Research Site, Sarasota, Florida
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Salt Lake City, Utah
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Valencia
- United Kingdom (5):
  - Research Site, Cambridge
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://breastcancerstudylocator.com/